CLINICAL TRIAL: NCT03536741
Title: The Role of Transversus Abdominis Plane Block and Rectus Sheath Block in Reduction of Postoperative Pain for Gynecological Benign Surgical Laparoscopic Procedures: a Randomized Controlled Trial
Brief Title: Role of TAP and RS Block in Reduction of Postoperative Pain for Gynecological Surgical Laparoscopic Procedures
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Corrado Terranova, Principal Investigator, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GIN-TAP 2017
Record Dates: First submitted 2018-03-09; First posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: TAP and RS Block
MeSH Terms: interventions — Anesthetics, Intravenous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALR (Experimental)
  Interventions: Procedure: TAP block and RS block + General Intravenous Anesthestic
- EV (Active Comparator)
  Interventions: Drug: General Intravenous Anesthetic

INTERVENTIONS:
Procedure: TAP block and RS block + General Intravenous Anesthestic — transversus abdominis plane block and rectus sheath block
  Arms: ALR
Drug: General Intravenous Anesthetic — General Intravenous Anesthetic
  Arms: EV

SUMMARY:
The present study aims to demonstrate the effectiveness of loco-regional wall anesthesia of the transversus abdominis plane block (TAP block) and the rectus sheath block (RS block), compared to intravenous analgesia, in terms of pain reduction, postoperative analgesic drugs consumption, patient satisfaction and decrease of LOS (length of stay), in patients undergoing benign gynecological laparoscopic surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing benign laparoscopic gynecological surgery
* age between 18 and 75 years
* BMI >18 e <35
* ECOG Performance Status 0-1

Exclusion Criteria:

* age < 18 or > 75 years
* BMI <18 or > 35
* ECOG Performance Status >1
* Allergy to local anesthetics
* Allergy to NSAIDs
* Chronic kidney failure > II class
* Systemic neoplastic disease actual or previous
* Actual pregnancy
* Active or recent pelvic inflammation
* Persistent coagulopathy
* Previous opioids consumption for chronic pain
* Neurological or cognitive disorders
* Conversion from laparoscopic to open surgery
* Onset of intraoperative complications

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-07-12 (Estimated); Study Completion 2018-07-12 (Estimated)

PRIMARY OUTCOMES:
postoperative pain in the first 72 hours after gynecological surgical procedures | postoperative pain in the first 72 hours after gynecological surgical procedures
  postoperative pain in the first 72 hours after gynecological surgical procedures
analgesic consumption in the first 72 hours after gynecological surgical procedures | analgesic consumption in the first 72 hours after gynecological surgical procedures
  analgesic consumption in the first 72 hours after gynecological surgical procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Campus Bio-medico, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No